CLINICAL TRIAL: NCT05432076
Title: Investigation of the Effect of Sleep Band and White Noise Use on Time to Sleep in Pediatric Intensive Care Patients Aged 3-12 Months
Brief Title: Sleep in Pediatric Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Ebru Kilic (Other)
Responsible Party: Sponsor-Investigator, Ebru Kilic, nurse, Cukurova University
Organization: Cukurova University (Other)
Other Study IDs: Çukurova Üniversitesi; 15619243304 (Other: çukurova üniversitesi)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Sleep
Keywords: White noise; sleep band; pediatric intensive care; baby/child

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: In the study, sleep bands and white noise will be used for sleep for the babies in the experimental group
  Interventions: Device: Sleep Band and White Noise
- control group: while the control group will not be interfered with

INTERVENTIONS:
Device: Sleep Band and White Noise — Not taking any sedative or anesthetic drug in the last 12 hours (Such duration of action) An average of 12 hours of sleepiness at the patient's departure and travel hindrance will.)
  * Being extubated
  * A Glasgow coma scale of 15 (to be investigated by the Glasgow coma scale).
  * Baby dreams of boredom
  * Besides pain (to the "Wong Baker Face Scale" used in the Pediatric Intensive Care Unit) evaluation).
  Other Names: Sleep Band; White Noise
  Groups: experimental group

SUMMARY:
This research will be carried out experimentally in order to investigate the Effect of Sleep Band and White Noise Use on the Time to Sleep in Pediatric Intensive Care Patients aged 3-12 months. The research will be carried out in Adana Province Seyhan State Hospital Pediatric Intensive Care Unit. The data obtained by creating experimental and control groups will be calculated. "Baby Information Form, Baby Sleep Problems Diagnosis Form, Baby Sleep Observation Form and Vital Findings Follow-up Chart" will be used to collect research data. In the study, sleep bands and white noise will be used for sleep for the babies in the experimental group, while the control group will not be interfered with. Ethics committee, institutional permission and informed consent from the parents of the infants will be obtained for the conduct of the study. SPSS demo package program will be used in data analysis. Examining the Effect Effect of Sleep Band and White Noise Use on Transition Time to Sleep in Pediatric Intensive Care Patients aged 3-12 months

, sleep ecology , sleep diagnostics Patients aged 3-12 months At the end of the research, it will be examined whether there is a difference between the sleep time, waking frequency and total sleep time of the babies in the experimental group using the sleep band and white noise, and the babies in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Not taking intravenous sedation and anesthetic drugs for the last 12 hours
* Extubated
* Infant patients who do not have respiratory distress
* Absence of pain

Exclusion Criteria:

* Mechanically ventilated and intubated patients
* Patients hospitalized with the diagnosis of respiratory distress
* Patients with vision and hearing problems

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample of the study consists of a total of 78 patients, 39 in the experimental and 39 in the control group. As a result of the power analysis using the G*Power 3.0.10 program; A total of at least 78 samples were found to be sufficient with 90% power and 5% margin of error (n1: 39, n2: 39).
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
sleep | 2 months
  This research will be carried out experimentally in order to investigate the Effect of Sleep Band and White Noise Use on the Time to Sleep in Pediatric Intensive Care Patients aged 3-12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Çetinkaya, Study Director — Cukurova University
Locations (1):
- Ebru Kaltar, Adana, Çukurova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided